CLINICAL TRIAL: NCT02558374
Title: A Double-masked, Randomized, Multi-center, Active-controlled, Parallel Group, 6-month Study With a 3-month Interim Analysis Assessing the Ocular Hypotensive Efficacy and Safety of AR-13324 Ophthalmic Solution, 0.02% QD Compared to Timolol Maleate Ophthalmic Solution, 0.5% BID in Patients With Elevated Intraocular Pressure
Brief Title: Double-masked Study of Netarsudil (AR-13324) Ophthalmic Solution in Subjects With Glaucoma or Ocular Hypertension
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Aerie Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AR-13324-CS304
Record Dates: First submitted 2015-09-16; First posted 2015-09-24 (Estimated); Results first posted 2018-04-06 (Actual); Last update posted 2018-04-06 (Actual); Status verified 2018-01

CONDITIONS: Open-angle Glaucoma; Ocular Hypertension
MeSH Terms: conditions — Glaucoma, Open-Angle; Ocular Hypertension | interventions — netarsudil; BID protein, human

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- AR-13324 Ophthalmic Solution 0.02% & placebo (Experimental): 1 drop AR-13324 in the evening (PM) & 1 drop placebo in the morning (AM) in both eyes (OU)
  Interventions: Drug: AR-13324 Ophthalmic Solution 0.02%; Other: Placebo
- Timolol Maleate Ophthalmic Solution 0.5% BID (Active Comparator): 1 drop twice daily (BID) in the morning (AM) & evening (PM) in both eyes (OU)
  Interventions: Drug: Timolol Maleate Ophthalmic Solution 0.5% BID

INTERVENTIONS:
Drug: AR-13324 Ophthalmic Solution 0.02% — 1 drop once daily (QD), PM, OU
  Other Names: Netarsudil
  Arms: AR-13324 Ophthalmic Solution 0.02% & placebo
Drug: Timolol Maleate Ophthalmic Solution 0.5% BID — 1 drop BID, AM/PM, OU
  Arms: Timolol Maleate Ophthalmic Solution 0.5% BID
Other: Placebo — 1 drop QD, AM, OU
  Arms: AR-13324 Ophthalmic Solution 0.02% & placebo

SUMMARY:
To evaluate ocular hypotensive efficacy and safety of Netarsudil (AR-13324) Ophthalmic Solution compared to Timolol Maleate Ophthalmic Solution.

ELIGIBILITY:
Inclusion Criteria:

1. 18 years of age or older
2. Diagnosis of open angle glaucoma or ocular hypertension in both eyes
3. Post-washout intraocular pressure >20mmHg and <30mmHg in 1 or both eyes at 2 qualification visits
4. Corrected visual acuity equivalent to 20/200
5. Able to give informed consent and follow study instructions

Exclusion Criteria:

1. Clinically significant ocular disease
2. Pseudoexfoliation or pigment dispersion component glaucoma, history of angle closure or narrow angles
3. Unmedicated intraocular pressure ≥30mmHg
4. Use of more than 2 ocular hypotensive medications within 30 days of screening
5. Known hypersensitivity to any component of the formulation
6. Previous glaucoma surgery or refractive surgery
7. Ocular trauma within 6 months prior to screening
8. Any ocular surgery or non-refractive laser treatment within 3 months prior to screening
9. Recent or current ocular infection or inflammation in either eye
10. Used ocular medication in either eye of any kind within 30 days of screening
11. Mean central corneal thickness >620µm at screening
12. Any abnormality preventing reliable applanation tonometry of either eye
13. Clinically significant abnormalities in lab tests at screening
14. Known hypersensitivity or contraindication to beta-adrenoceptor antagonists
15. Clinically significant systemic disease
16. Participation in any investigational study within 60 days prior to screening
17. Used any systemic medication that could have a substantial effect in intraocular pressure within 30 days prior to screening
18. Women who are pregnant, nursing, planning a pregnancy or not using a medically acceptable form of birth control

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 708 (Actual)
Dates: Start 2015-09; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Theresa Heah, MD, Study Director — Aerie Pharmaceuticals, Inc
Locations (1):
- Aerie Pharmaceuticals, Bedminster, New Jersey, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited at 53 sites starting in September 2015
Groups:
- Timolol Maleate Ophthalmic Solution 0.5% BID: 1 drop twice daily (BID) in the morning (AM) and evening (PM) in both eyes (OU)
Period: Overall Study
Arm/Group | AR-13324 Ophthalmic Solution 0.02% & Placebo | Timolol Maleate Ophthalmic Solution 0.5% BID
Started | 351 | 357
Completed | 243 | 314
Not Completed | 108 | 43

BASELINE CHARACTERISTICS:
Groups:
- AR-13324 Ophthalmic Solution 0.02% & Placebo: 1 drop AR-13324 in the evening (PM) and 1 drop placebo in the morning (AM) in both eyes (OU)
- Total: Total of all reporting groups
Arm/Group | AR-13324 Ophthalmic Solution 0.02% & Placebo | Timolol Maleate Ophthalmic Solution 0.5% BID | Total
Number analyzed (Participants) | 351 | 357 | 708
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.1 (11.55) | 64.5 (10.97) | 64.3 (11.25)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 208 | 237 | 445
  Male | 143 | 120 | 263
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 89 | 87 | 176
  Not Hispanic or Latino | 262 | 270 | 532
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 7 | 6 | 13
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 84 | 75 | 159
  White | 259 | 274 | 533
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: IOP (Intraocular Pressure)
Description: The primary efficacy outcome is mean IOP
Time Frame: 3 months
Population: Per-Protocol Population
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | AR-13324 Ophthalmic Solution 0.02% & Placebo | Timolol Maleate Ophthalmic Solution 0.5% BID
Number analyzed (Participants) | 306 | 316
mmHg
  Day 1, 0800 hours | 23.93 (2.441) | 23.89 (2.318)
  Day 1, 1000 hours | 22.67 (2.826) | 22.77 (2.565)
  Day 1, 1600 hours | 22.17 (2.857) | 22.04 (2.708)
  Day 15, 0800 hours | 19.20 (3.833) | 18.60 (3.396)
  Day 15, 1000 hours | 17.93 (3.678) | 17.80 (3.237)
  Day 15, 1600 hours | 17.76 (3.527) | 17.85 (3.102)
  Day 43, 0800 hours | 19.45 (3.929) | 18.52 (3.316)
  Day 43, 1000 hours | 18.12 (3.560) | 17.89 (3.157)
  Day 43, 1600 hours | 17.89 (3.438) | 17.88 (3.356)
  Day 90, 0800 hours | 19.24 (3.889) | 18.35 (3.196)
  Day 90, 1000 hours | 18.30 (3.637) | 17.60 (3.173)
  Day 90, 1600 hours | 18.02 (3.644) | 17.66 (3.080)

2. Secondary Outcome: Extent of Exposure
Description: Exposure to study medication in days for all treatment groups
Time Frame: 6 months
Population: Safety Population
Measure: Mean (Standard Deviation); unit: days
Arm/Group | AR-13324 Ophthalmic Solution 0.02% & Placebo | Timolol Maleate Ophthalmic Solution 0.5% BID
Number analyzed (Participants) | 351 | 357
days | 147.4 (54.47) | 167.7 (36.40)

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | AR-13324 Ophthalmic Solution 0.02% & Placebo | Timolol Maleate Ophthalmic Solution 0.5% BID
All-Cause Mortality (participants affected / at risk) | 1/351 | 0/357
Serious Adverse Events (participants affected / at risk) | 8/351 | 10/357
Other Adverse Events (participants affected / at risk) | 245/351 | 139/357
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | AR-13324 Ophthalmic Solution 0.02% & Placebo (N=351) | Timolol Maleate Ophthalmic Solution 0.5% BID (N=357)
Bladder Cancer Recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Chronic Myeloid Leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Invasive Ductal Breast Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Papillary Thyroid Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Uterine Leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Atrial Fibrillation (Cardiac disorders) | 0 | 1
Cardiac Arrest (Cardiac disorders) | 1 | 0
Cardiomegaly (Cardiac disorders) | 0 | 1
Coronary Artery Disease (Cardiac disorders) | 0 | 1
Myocardial Infarction (Cardiac disorders) | 1 | 0
Transient Ischaemic Attack (Nervous system disorders) | 1 | 1
Facial Paralysis (Nervous system disorders) | 0 | 1
Abdominal Discomfort (Gastrointestinal disorders) | 0 | 1
Gastric Volvulus (Gastrointestinal disorders) | 1 | 0
Hiatus Hernia (Gastrointestinal disorders) | 1 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 1
Radius Fracture (Injury, poisoning and procedural complications) | 0 | 1
Pneumonia (Infections and infestations) | 0 | 1
Mental Status Changes (Psychiatric disorders) | 0 | 1
Bladder Prolapse (Renal and urinary disorders) | 1 | 0
Cervical Dysplasia (Reproductive system and breast disorders) | 1 | 0
Pneumonia Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | AR-13324 Ophthalmic Solution 0.02% & Placebo (N=351) | Timolol Maleate Ophthalmic Solution 0.5% BID (N=357)
Conjunctival Hyperaemia (Eye disorders) | 168 | 33
Cornea Verticillata (Eye disorders) | 86 | 0
Conjunctival Haemorrhage (Eye disorders) | 56 | 11
Lacrimation Increased (Eye disorders) | 26 | 5
Erythema of Eyelid (Eye disorders) | 26 | 2
Vision Blurred (Eye disorders) | 22 | 4
Instillation Site Pain (General disorders) | 83 | 92
Instillation Site Erythema (General disorders) | 36 | 4
Vital Dye Staining Cornea Present (Investigations) | 34 | 24

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No